CLINICAL TRIAL: NCT02344888
Title: Adding Prednisolone During Ovulation Induction With Clomiphene Citrate in Lean Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome
Brief Title: Adding Prednisolone During Ovulation Induction With CC in Lean Women With CC Resistant PCOS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahmoud Thabet (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Thabet, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMA1
Record Dates: First submitted 2015-01-18; First posted 2015-01-26 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Infertility; Polycystic Ovarian Syndrome
Keywords: PCOS; Clomiphene citrate resistant; Prednisolone
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Clomiphene; Prednisolone; Methylprednisolone; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomiphene citrate-Prednisolone group (Active Comparator): Women will receive clomiphene citrate and prednisolone
  Interventions: Drug: Clomiphene citrate and Prednisolone
- Clomiphene citrate-placebo group (Active Comparator): Women will receive clomiphene citrate and folic acid 0.5mg (placebo)
  Interventions: Drug: Clomiphene citrate and folic acid

INTERVENTIONS:
Drug: Clomiphene citrate and Prednisolone — Women will receive clomiphene citrate (150 mg/day for 5 consecutive days from day 2 of the cycle) and prednisolone (5 mg/day for 10 consecutive days from day 2 of the cycle)
  Other Names: Clomid and Hostacortin-H
  Arms: Clomiphene citrate-Prednisolone group
Drug: Clomiphene citrate and folic acid — Women will receive clomiphene citrate alone (150 mg/day for 5 consecutive days from day 2 of the cycle) and folic acid (0.5 mg/day for 10 consecutive days from day 2 of the cycle)
  Other Names: Clomid and folic acid
  Arms: Clomiphene citrate-placebo group

SUMMARY:
The purpose of this study is to evaluate the effect of concomitant administration of prednisolone during use of clomiphene citrate (CC) for induction of ovulation in infertile lean women having CC resistant polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; CC-Prednisolone group and CC-placebo group. Women in the CC-Prednisolone group will receive CC (150 mg/day for 5 consecutive days from day 2 of the cycle) and prednisolone tablet (5 mg/day for 10 consecutive days from day 2 of the cycle). Women in the CC-placebo group will receive CC alone (150 mg/day for 5 consecutive days from day 2 of the cycle) and folic acid tablet (0.5 mg/day for 10 consecutive days from day 2 of the cycle). Transvaginal sonography (TVS) scan will be performed regularly for monitoring of follicular growth (folliculometry); starting from day 10 of the stimulation cycle and repeated every 2-3 days. When there will be at least one follicle ≥ 18 mm in diameter, final oocyte maturation will be induced by intramuscular administration of 10000 IU of human chorionic gonadotropin (HCG) and timed intercourse will be advised. If there will be no follicle ≥ 12 mm by day 16 of the cycle, monitoring of follicular growth will be discontinued and the cycle will be presumed to be anovulatory. Ovulation will be documented by TVS scan one week after triggering of oocyte maturation and will be confirmed by assessing the mid-luteal serum progesterone level. Each woman will be subjected to ovarian stimulation for a maximum of 3 consecutive cycles except if she gets pregnant in the first or second cycle

ELIGIBILITY:
Inclusion Criteria:

* Infertile lean women with PCOS as defined by the Rotterdam criteria.
* CC resistance (defined as failure of ovulation after receiving 150 mg/day of CC for 5 consecutive days per cycle, for at least 3 consecutive cycles).

Exclusion Criteria:

* Age < 20 or > 35 years.
* Body mass index (BMI) < 18.5 kg/m2 or > 25 kg/m2.
* Presence of any infertility factor other than anovulatory PCOS.
* Previous history of ovarian surgery or surgical removal of one ovary.
* Previous exposure to cytotoxic drugs or pelvic irradiation.
* Oral hypoglycemic or hormonal therapy either currently or in the preceding 3 months.
* Metabolic or hormonal abnormalities

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Ovulation rate | 3 months
  Number of ovulatory cycles divided by the number of stimulation cycles

SECONDARY OUTCOMES:
Number of ovarian follicles ≥ 18 mm on day of HCG administration | 3 months
  Number of ovarian follicles ≥ 18 mm by TVS on day of HCG administration
Endometrial thickness on day of HCG administration | 3 months
  Endometrial thickness by TVS on day of HCG administration
Clinical pregnancy rate | 6-8 weeks gestational age
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 6-8 weeks gestational age) divided by the number of women

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Abdelrazik, Dr, Principal Investigator — Mansoura University; Mahmoud Thabet, D, Study Director — Mansoura University
Locations (2):
- Egypt (2):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided